CLINICAL TRIAL: NCT05870943
Title: Hybrid Argon Plasma Coagulation and Endoscopic Sleeve Gastroplasty Trial: A Single-Center Randomized Controlled Validation Trial in a Community Setting
Brief Title: Hybrid Argon Plasma Coagulation and Endoscopic Sleeve Gastroplasty Validation Study
Acronym: HAPCET2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: True You Weight Loss (Other)
Collaborators: Erbe USA Incorporated (Other); Erbe Elektromedizin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCT-001
Record Dates: First submitted 2023-04-24; First posted 2023-05-23 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: 1:1 allocation to experimental and control group using variable block randomization
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and care providers will be blinded to the results of randomization. They will remain blinded until the end of the study, or if there is a medical or surgical safety concern.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Argon Plasma Coagulation and Endoscopic Sleeve Gastroplasty (Experimental): Hybrid APC will be utilized to first ablate the gastric mucosa along the greater curve of the stomach, followed immediately by endoscopic full-thickness tissue acquisition and plication using 2-0 Prolene synthetic sutures via the Apollo ESG platform.
  Interventions: Procedure: Hybrid Argon Plasma Coagulation; Procedure: Endoscopic Sleeve Gastroplasty
- Endoscopic Sleeve Gastroplasty (Active Comparator): Endoscopic full-thickness tissue acquisition and plication using 2-0 Prolene synthetic sutures via the Apollo ESG platform.
  Interventions: Procedure: Endoscopic Sleeve Gastroplasty

INTERVENTIONS:
Procedure: Hybrid Argon Plasma Coagulation — Hybrid APC will be utilized to first ablate the gastric mucosa along the greater curve of the stomach.
  Arms: Hybrid Argon Plasma Coagulation and Endoscopic Sleeve Gastroplasty
Procedure: Endoscopic Sleeve Gastroplasty — Endoscopic full-thickness tissue acquisition and plication using 2-0 Prolene synthetic sutures via the Apollo ESG platform.

SUMMARY:
The purpose of this research is to evaluate the clinical safety, durability, and weight loss outcomes of the hybrid argon plasma coagulation + endoscopic sleeve gastroplasty (HAPC-ESG) procedure when compared to traditional endoscopic sleeve gastroplasty (ESG) alone. ESG was proven to be feasible in human subjects in 2013 and since then has become the most commonly performed endoscopic bariatric remodeling procedure. However, this procedure may be enhanced with the addition of the hybrid argon plasma coagulation (HAPC) technique, leading to enhanced weight loss, durability, and metabolic benefits. Argon plasma coagulation (APC) is a method of non-contact thermal hemostasis initially created to assist in inducing hemostasis utilizing a high-frequency current to the targeted area. This is a validation study of a pilot randomized control trial which will evaluate the safety, durability, and effects on weight loss of the combined HAPC-ESG approach when compared to traditional ESG alone.

DETAILED DESCRIPTION:
Obesity is a chronic disease state driven by the imbalance of caloric intake and expenditure and mediated by multiple central and peripheral pathways that may serve as targets for therapeutic interventions. The endoscopic sleeve gastroplasty (ESG) is a per oral gastric remodeling technique that employs full-thickness suturing to imbricate the stomach along the greater curvature to achieve a restricted, sleeve-like configuration. Argon Plasma Coagulation (APC) is a method of non-contact thermal hemostasis which utilizes a high-frequency current applied to the target tissue through an argon plasma jet to induce hemostasis and a homogenous surface coagulation with a limited depth of penetration. APC is a widely used therapy in the luminal digestive tract to provide non-contact, targeted thermal injury for mucosal ablation and may therefore allow for a greater submucosal component of healing between tissue plications and, consequently, greater durability of the gastroplasty. Enhanced fibrosis along the site of endoscopic plications with the addition of APC could decrease the incidence of weight regain in patients undergoing ESG and capitalize on the metabolic benefits of gastric mucosal revitalization reported with APC alone. In this study, the investigators propose to evaluate the durability of endoscopic plications, weight loss outcomes, and improvements in obesity related co-morbidities for the combined hybrid argon plasma coagulation plus endoscopic sleeve gastroplasty (HAPC-ESG) procedure when compared to traditional ESG. Investigators hypothesize that HAPC-ESG will provide greater durability of the gastroplasty construct than traditional ESG. This is a single-center, randomized, single-blinded clinical trial evaluating the efficacy and safety of HAPC-ESG for weight loss and improvement in obesity-related co-morbidities compared to ESG alone. The study population includes adult patients who are seeking ESG at True You Weight Loss in Cary, NC with a BMI ≥ 30 and ≤40 kg/m² who have failed to achieve and maintain weight loss with a non-surgical management.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65
2. BMI ≥ 30 and ≤40 kg/m²
3. Willingness to comply with the substantial lifelong dietary restrictions required by the procedure.
4. History of failure with non-surgical weight-loss methods.
5. Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing laboratory tests, and completing diet counseling.
6. Residing within a reasonable driving distance from the investigator's office (Cary, NC) and able to travel to the investigator to complete all routine follow-up visits as applicable
7. Ability to give informed consent.
8. Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods.
9. Reliable access to wi-fi and/or internet services.

Exclusion Criteria:

1. History of foregut or gastrointestinal (GI) surgery (except uncomplicated cholecystectomy or appendectomy).
2. Prior gastrointestinal surgery with sequelae, i.e., obstruction, and/or adhesive peritonitis or known abdominal adhesions.
3. Prior open or laparoscopic bariatric surgery.
4. Prior surgery of any kind on the esophagus, stomach, or any type of hiatal hernia surgery.
5. Any inflammatory disease of the gastrointestinal tract including severe (LA Grade C or D) esophagitis, Barrett's esophagus, gastric ulceration, duodenal ulceration, cancer, or specific inflammatory disease such as Crohn's disease or celiac disease.
6. Potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresias or stenoses.
7. Gastrointestinal stromal tumors, history of premalignant gastric lesions (intestinal metaplasia), history of familial and nan-familial adenomatous syndromes.
8. A gastric mass or gastric polyps > 1 cm in size.
9. A hiatal hernia > 4cm of axial displacement of the z-line above the diaphragm or severe or intractable gastro-esophageal reflux symptoms.
10. A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the endoscope.
11. Achalasia or any other severe esophageal motility disorder
12. Severe coagulopathy.
13. Insulin-dependent diabetes (either Type 1 or Type 2) or a significant likelihood of requiring insulin treatment in the following 12 months or a HgbA1C≥9.
14. Subjects with any serious health condition unrelated to their weight that would increase the risk of endoscopy.
15. Chronic abdominal pain.
16. Motility disorders of the GI tract such as gross esophageal motility disorders, gastroparesis or intractable constipation.
17. Hepatic insufficiency or cirrhosis.
18. Use of an intragastric device prior to this study due to the increased thickness of the stomach wall preventing effective suturing.
19. Active psychological issues preventing participation in a life-style modification program as determined by a psychologist.
20. Patients unwilling to participate in an established medically supervised diet and behavior modification program, with routine medical follow-up.
21. Patients receiving daily prescribed treatment with high dose aspirin (> 81mg daily), anti-inflammatory agents, anticoagulants, or other gastric irritants.
22. Patients who are unable or unwilling to take prescribed proton pump inhibitor medication.
23. Patients who are pregnant or breast-feeding.
24. Patients currently taking weight-loss medications or other therapies for weight loss within the prior 6 months.
25. Subjects with severe cardiopulmonary disease or other serious organic disease which might include known history of coronary artery disease, myocardial infarction within the past 6 months, poorly controlled hypertension, required use of NSAIDs.
26. Subjects taking medications on specified hourly intervals that may be affected by changes to gastric emptying, such as anti-seizure or anti-arrhythmic medications.
27. Subjects who are taking corticosteroids, immunosuppressants, and narcotics.
28. Symptomatic congestive heart failure, cardiac arrhythmia, or unstable coronary artery disease.
29. Pre-existing respiratory disease such as moderate or severe chronic obstructive pulmonary disease (COPD) requiring steroids, pneumonia, or cancer.
30. Diagnosis of autoimmune connective tissue disorder (e.g. Systemic lupus erythematosus, scleroderma) or immunocompromised.
31. Specific diagnosed genetic disorder such as Prader Willi syndrome.
32. Eating disorders including night eating syndrome (NES), bulimia, binge eating disorder, or compulsive overeating.
33. Known history of endocrine disorders affecting weight such as uncontrolled hypothyroidism.
34. At the discretion of the PI for subject safety
35. If minority inclusion population target of 10% has not been reached by the 90% enrollment mark (example 43 of 48 subjects), the remaining enrollments will be reserved for minority subjects (example 5 of 48 subjects).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Durability assessed by blinded physician(s) with expertise in endoscopic sleeve gastroplasty (ESG) procedures graded according to a priori standardized criteria. | 6 Months
  The primary outcomes are durability of plications and endoscopic sutures on repeat endoscopy at 6 months, in the two randomized arms. Durability of plications and endoscopic sutures will be assessed by blinded physician(s) with expertise in ESG who will assess sleeve-like anatomy (scale: None, Some, Typical), tissue bonding (scale: None, Some, Plenty), and tightness of sutures (scale: Loose, Somewhat tight, Tight) to measure durability.

SECONDARY OUTCOMES:
%TBWL | 6 Month
  Compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis
%EWL | 6 and 12 month
  Compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis
Blood Pressure | 6 month
  Systolic and diastolic blood pressure compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis
HbA1c percentage | 6 Month
  Percentage of red blood cells that have glucose-coated hemoglobin compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis
Change in quality of life measured by Questionnaire: Short Form Health Survey (SF-36) | 6 Month
  Changes in Short Form Health Survey responses compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis. Minimum score of 38 and maximum score of 149. Quality of life outcome determined by changes in individual scores on each respective question.
Change in quality of life measured by Questionnaire: Impact of Weight on Quality of Life-Lite (IWQOL-Lite) | 6 Month
  Changes in Impact of Weight on Quality of Life-Lite responses compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis. Minimum score of 31 and maximum score of 155 with a higher score reflective of poor self-assessed quality of life.
Change in depression measured by Questionnaire: Patient Health Questionnaire (PHQ-9) | 6 Month
  Changes in Patient Health Questionnaire (PHQ-9) responses compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis. Minimum score of 0 and maximum score of 27 with lower scores reflective of no or mild depression, medium scores reflective of moderate depression, and high scores reflective of severe depression.
Change in eating behavior measured by Questionnaire: The Three-Factor Eating Questionnaire (TFEQ-r18) | 6 Month
  Change in eating behaviors measured by Questionnaire: The Three-Factor Eating Questionnaire (TFEQ-r18) compared between treatment arms using ANCOVA with adjustment for the same variables specified in the primary analysis. Minimum score of 18 and maximum score of 80 with higher scores associated with disinhibition, hunger, and decreased cognitive restraint.
Binary Outcomes: ≥25% change in %EWL | 6 Month
  Compared between treatment arms by Pearson Chi-square test.
Incidence of esophagitis | 6 Month
  Incidence of esophagitis identified by trained physician(s) to be compared between treatment arms by Pearson Chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E McGowan, MD, MSCR, Principal Investigator — CEO/Medical Director
Locations (1):
- True You Weight Loss, Cary, North Carolina, United States

REFERENCES:
- [Background] Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of Obesity and Severe Obesity Among Adults: United States, 2017-2018. NCHS Data Brief. 2020 Feb;(360):1-8. PMID 32487284
- [Background] Ward ZJ, Bleich SN, Cradock AL, Barrett JL, Giles CM, Flax C, Long MW, Gortmaker SL. Projected U.S. State-Level Prevalence of Adult Obesity and Severe Obesity. N Engl J Med. 2019 Dec 19;381(25):2440-2450. doi: 10.1056/NEJMsa1909301. PMID 31851800
- [Background] Flegal KM, Kit BK, Orpana H, Graubard BI. Association of all-cause mortality with overweight and obesity using standard body mass index categories: a systematic review and meta-analysis. JAMA. 2013 Jan 2;309(1):71-82. doi: 10.1001/jama.2012.113905. PMID 23280227
- [Background] Adams KF, Schatzkin A, Harris TB, Kipnis V, Mouw T, Ballard-Barbash R, Hollenbeck A, Leitzmann MF. Overweight, obesity, and mortality in a large prospective cohort of persons 50 to 71 years old. N Engl J Med. 2006 Aug 24;355(8):763-78. doi: 10.1056/NEJMoa055643. Epub 2006 Aug 22. PMID 16926275
- [Background] Prospective Studies Collaboration; Whitlock G, Lewington S, Sherliker P, Clarke R, Emberson J, Halsey J, Qizilbash N, Collins R, Peto R. Body-mass index and cause-specific mortality in 900 000 adults: collaborative analyses of 57 prospective studies. Lancet. 2009 Mar 28;373(9669):1083-96. doi: 10.1016/S0140-6736(09)60318-4. Epub 2009 Mar 18. PMID 19299006
- [Background] Wadden TA, Butryn ML, Wilson C. Lifestyle modification for the management of obesity. Gastroenterology. 2007 May;132(6):2226-38. doi: 10.1053/j.gastro.2007.03.051. PMID 17498514
- [Background] Kheniser K, Saxon DR, Kashyap SR. Long-Term Weight Loss Strategies for Obesity. J Clin Endocrinol Metab. 2021 Jun 16;106(7):1854-1866. doi: 10.1210/clinem/dgab091. PMID 33595666
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- [Background] Wadden TA, Bailey TS, Billings LK, Davies M, Frias JP, Koroleva A, Lingvay I, O'Neil PM, Rubino DM, Skovgaard D, Wallenstein SOR, Garvey WT; STEP 3 Investigators. Effect of Subcutaneous Semaglutide vs Placebo as an Adjunct to Intensive Behavioral Therapy on Body Weight in Adults With Overweight or Obesity: The STEP 3 Randomized Clinical Trial. JAMA. 2021 Apr 13;325(14):1403-1413. doi: 10.1001/jama.2021.1831. PMID 33625476
- [Background] Davies M, Faerch L, Jeppesen OK, Pakseresht A, Pedersen SD, Perreault L, Rosenstock J, Shimomura I, Viljoen A, Wadden TA, Lingvay I; STEP 2 Study Group. Semaglutide 2.4 mg once a week in adults with overweight or obesity, and type 2 diabetes (STEP 2): a randomised, double-blind, double-dummy, placebo-controlled, phase 3 trial. Lancet. 2021 Mar 13;397(10278):971-984. doi: 10.1016/S0140-6736(21)00213-0. Epub 2021 Mar 2. PMID 33667417
- [Background] Enebo LB, Berthelsen KK, Kankam M, Lund MT, Rubino DM, Satylganova A, Lau DCW. Safety, tolerability, pharmacokinetics, and pharmacodynamics of concomitant administration of multiple doses of cagrilintide with semaglutide 2.4 mg for weight management: a randomised, controlled, phase 1b trial. Lancet. 2021 May 8;397(10286):1736-1748. doi: 10.1016/S0140-6736(21)00845-X. Epub 2021 Apr 22. PMID 33894838
- [Background] Bal BS, Finelli FC, Shope TR, Koch TR. Nutritional deficiencies after bariatric surgery. Nat Rev Endocrinol. 2012 Sep;8(9):544-56. doi: 10.1038/nrendo.2012.48. Epub 2012 Apr 24. PMID 22525731
- [Background] Proietto J. Why is treating obesity so difficult? Justification for the role of bariatric surgery. Med J Aust. 2011 Aug 1;195(3):144-6. doi: 10.5694/j.1326-5377.2011.tb03242.x. PMID 21806533
- [Background] Hedjoudje A, Abu Dayyeh BK, Cheskin LJ, Adam A, Neto MG, Badurdeen D, Morales JG, Sartoretto A, Nava GL, Vargas E, Sui Z, Fayad L, Farha J, Khashab MA, Kalloo AN, Alqahtani AR, Thompson CC, Kumbhari V. Efficacy and Safety of Endoscopic Sleeve Gastroplasty: A Systematic Review and Meta-Analysis. Clin Gastroenterol Hepatol. 2020 May;18(5):1043-1053.e4. doi: 10.1016/j.cgh.2019.08.022. Epub 2019 Aug 20. PMID 31442601
- [Background] Sharaiha RZ, Hajifathalian K, Kumar R, Saunders K, Mehta A, Ang B, Skaf D, Shah S, Herr A, Igel L, Dawod Q, Dawod E, Sampath K, Carr-Locke D, Brown R, Cohen D, Dannenberg AJ, Mahadev S, Shukla A, Aronne LJ. Five-Year Outcomes of Endoscopic Sleeve Gastroplasty for the Treatment of Obesity. Clin Gastroenterol Hepatol. 2021 May;19(5):1051-1057.e2. doi: 10.1016/j.cgh.2020.09.055. Epub 2020 Oct 1. PMID 33011292
- [Background] Mahmoud T, Vargas EJ, Ghazi R, Abusaleh R, Storm AC, Abu Dayyeh BK. The Osculating Circles Gastroplasty: A Novel Endoscopic Submucosal Resection Enhanced Endoluminal Suturing for Obesity. Gastroenterology. 2021 Dec;161(6):1806-1808.e1. doi: 10.1053/j.gastro.2021.08.059. Epub 2021 Sep 26. No abstract available. PMID 34587488
- [Background] Zenker M. Argon plasma coagulation. GMS Krankenhhyg Interdiszip. 2008 Nov 3;3(1):Doc15. PMID 20204117
- [Background] Jirapinyo P, de Moura DTH, Dong WY, Farias G, Thompson CC. Dose response for argon plasma coagulation in the treatment of weight regain after Roux-en-Y gastric bypass. Gastrointest Endosc. 2020 May;91(5):1078-1084. doi: 10.1016/j.gie.2019.12.036. Epub 2020 Jan 3. PMID 31904378
- [Background] Itani MI, Farha J, Sartoretto A, Abbarh S, Badurdeen D, de Moura DTH, Kumbhari V. Endoscopic sleeve gastroplasty with argon plasma coagulation: A novel technique. J Dig Dis. 2020 Nov;21(11):664-667. doi: 10.1111/1751-2980.12939. PMID 32916766
- [Background] Lee JH, Johannes RS, Van Dam J, et al. 7087 Argon plasma coagulation in endoscopic therapy. Gastrointestinal Endoscopy 2000;51:AB264.
- [Background] Mitchell NS, Catenacci VA, Wyatt HR, Hill JO. Obesity: overview of an epidemic. Psychiatr Clin North Am. 2011 Dec;34(4):717-32. doi: 10.1016/j.psc.2011.08.005. PMID 22098799
- [Background] Abu Dayyeh BK, Rajan E, Gostout CJ. Endoscopic sleeve gastroplasty: a potential endoscopic alternative to surgical sleeve gastrectomy for treatment of obesity. Gastrointest Endosc. 2013 Sep;78(3):530-5. doi: 10.1016/j.gie.2013.04.197. Epub 2013 May 24. PMID 23711556
- [Background] Marchesini SD, Baretta GA, Cambi MP, Marchesini JB. Endoscopic plasma argon coagulation in treatment of weight regain after bariatric surgery: what does the patient think about this? Arq Bras Cir Dig. 2014;27 Suppl 1(Suppl 1):47-50. doi: 10.1590/s0102-6720201400s100012. PMID 25409966
- [Background] Dhindsa BS, Saghir SM, Naga Y, Dhaliwal A, Ramai D, Cross C, Singh S, Bhat I, Adler DG. Efficacy of transoral outlet reduction in Roux-en-Y gastric bypass patients to promote weight loss: a systematic review and meta-analysis. Endosc Int Open. 2020 Oct;8(10):E1332-E1340. doi: 10.1055/a-1214-5822. Epub 2020 Sep 22. PMID 33015335
- [Background] Storm AC, Thompson CC. Endoscopic Treatments Following Bariatric Surgery. Gastrointest Endosc Clin N Am. 2017 Apr;27(2):233-244. doi: 10.1016/j.giec.2016.12.007. PMID 28292402
- [Background] Jaruvongvanich V, Vantanasiri K, Laoveeravat P, Matar RH, Vargas EJ, Maselli DB, Alkhatry M, Fayad L, Kumbhari V, Fittipaldi-Fernandez RJ, Hollenbach M, Watson RR, Gustavo de Quadros L, Galvao Neto M, Aepli P, Staudenmann D, Brunaldi VO, Storm AC, Martin JA, Gomez V, Abu Dayyeh BK. Endoscopic full-thickness suturing plus argon plasma mucosal coagulation versus argon plasma mucosal coagulation alone for weight regain after gastric bypass: a systematic review and meta-analysis. Gastrointest Endosc. 2020 Dec;92(6):1164-1175.e6. doi: 10.1016/j.gie.2020.07.013. Epub 2020 Jul 18. PMID 32692991
- [Background] Catalano MF, Rudic G, Anderson AJ, Chua TY. Weight gain after bariatric surgery as a result of a large gastric stoma: endotherapy with sodium morrhuate may prevent the need for surgical revision. Gastrointest Endosc. 2007 Aug;66(2):240-5. doi: 10.1016/j.gie.2006.06.061. Epub 2007 Feb 28. PMID 17331511
- [Background] Baretta GA, Alhinho HC, Matias JE, Marchesini JB, de Lima JH, Empinotti C, Campos JM. Argon plasma coagulation of gastrojejunal anastomosis for weight regain after gastric bypass. Obes Surg. 2015 Jan;25(1):72-9. doi: 10.1007/s11695-014-1363-2. PMID 25005812
- [Background] de Moura DTH, Badurdeen DS, Ribeiro IB, Leite EFMDSD, Thompson CC, Kumbhari V. Perspectives toward minimizing the adverse events of endoscopic sleeve gastroplasty. Gastrointest Endosc. 2020 Nov;92(5):1115-1121. doi: 10.1016/j.gie.2020.06.038. Epub 2020 Jun 17. No abstract available. PMID 32562607